CLINICAL TRIAL: NCT06918977
Title: Evaluation of a Novel Telemedicine Clinic for Patients With DM2 on Multiple Daily Insulin (MDI) Regimens
Brief Title: Improving Glycemic Control With Telemedicine and Smart Insulin Pens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00113553
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; CGM device; Smart Insulin Pen
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Group (Experimental): Intervention group: will be managed with telehealth and InPen Smart insulin pens
  Interventions: Device: InPen Smart insulin pen
- Control Group (Other): Control group: will be managed by telehealth and the traditional/standard insulin pen (widely used)
  Interventions: Other: traditional/standard insulin pen

INTERVENTIONS:
Device: InPen Smart insulin pen — InPen is a reusable pen injector which allows the user to dial the desired dose of insulin to be administered. The dose calculator a component of the InPen app calculates an insulin dose or carbohydrate intake based on user entered data. Prior to use, the patient -specific target blood glucose, insulin-to-carbohydrate ratio, and insulin sensitivity parameters are to be programmed into the software.
  Arms: Intervention Group
Other: traditional/standard insulin pen — personal prescribed insulin pen
  Arms: Control Group

SUMMARY:
Almost 40% of veterans have diabetes, the proposed research may improve clinical care among veterans with diabetes. In this application we are going to examine whether utilizing Smart Insulin pens (SIPs) with CGMs and telemedicine is a better tool for managing diabetes compared to traditional insulin pens, CGMs and telemedicine, leading to improved blood sugar control and better clinical outcomes.

DETAILED DESCRIPTION:
Diabetes is affecting millions of Americans. High glucose levels lead to complications such as heart attacks, stroke or blindness. Reducing high glucose levels may unfortunately lead to very low glucose values-hypoglycemia, a condition that can lead to loss of consciousness or even death. Both of these conditions, high and low glucose levels, can therefore lead to visits to the Emergency department or hospitalizations. In fact, patients with diabetes have frequent admissions to the hospital. Additionally, many of them are admitted again, immediately or in less than 30 days after hospital discharge.

Most patients with diabetes are monitoring their glucose values with finger-stick glucose testing. Continuous Glucose Monitors (CGM)s are new devices that can monitor glucose continuously (every couple of minutes) without the need of finger-stick glucose testing. Similar to the glucometers, CGM devices can record glucose values, which can then be obtained by the clinicians, who can help them to modify DM medications.

In addition to using CGM devices for diabetes management, smart insulin pens can be used in order to help with diabetes control. These devices can store and transfer data to the medical doctors, making them aware about the patients' glucose values.

Moreover there are different health solutions available to manage patients including mobile health and telemedicine, which can help combining and transferring these data remotely. Briefly, telemedicine is a way to deliver healthcare where providers and patients communicate through alternative methods ( for example, telephone or other electronic method) instead of traditional in-person office visits. Using telemedicine to replace some routine office visits can improve access to healthcare.

Subjects will be randomly assigned in 2 groups: One group will include patients with SIPs, CGMs and telemedicine and the other group will use traditional insulin pens, CGMs and telemedicine

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* MDI insulin treated (receiving MDI for at least 3 months prior to the study)

Exclusion Criteria:

* DM patients not treated with MDI for at least 3 months (i.e diet only, any combination of non-insulin antidiabetic drugs only, basal insulin only or bolus/short acting insulin only)
* Patients with DM at the time of screening on insulin pumps
* Pregnant patients
* Patients with extensive skin disease or allergies that preclude wearing the CGM sensor
* Patients who have end-stage renal disease requiring dialysis
* Patients with significant psychiatric illness or any other condition rendering the subject incapable of understanding the objectives and potential consequences of the study
* Patients who receive hydroxyurea or who are on long (chronic) treatment with acetaminophen
* Patients who were started on non-insulin DM medications or had a dose change within 60 days or less prior to study participation
* Patient does not have or not able to gain access to a smartphone which is compatible with the necessary applications for DAT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in hyperglycemia | 3 months
  This will be evaluated by decrease HbA1c

SECONDARY OUTCOMES:
Change in hyperglycemia | 6 months
  This will be evaluated by decrease in HbA1c

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baltimore VA Maryland Center, Baltimore, Maryland
  - VAMHCS, Diabetes Outpatient Clinic, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided